CLINICAL TRIAL: NCT03285958
Title: Promoting Physical Activity for Chronic Pain Management Among Older Adults in Detroit: Comparing Technology-Based Strategies
Brief Title: Tracking Physical Activity for Chronic Pain Management Among Older Adults in Detroit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mary Janevic, Assistant Research Scientist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00133021
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEPS Intervention Group (Experimental): Participants will receive a wearable physical activity monitor and will be asked to report their daily step count in 3 different ways (2 weeks each of SMS text messages, Interactive Voice Response calls (IVR), automatic upload) during the 6-week study period.
  Interventions: Behavioral: STEPS Intervention
- STEPS Control Group (No Intervention): Participants in this group will not receive a wearable physical activity monitor and will not be asked to report their step count.

INTERVENTIONS:
Behavioral: STEPS Intervention — Participants in the STEPS (Seniors Tracking Exercise for Pain Self-management) intervention will receive a commercially-available, wearable physical activity monitor. They will be asked to wear this monitor during waking hours for 6 weeks, reporting their daily step count every evening. The way in which participants report steps will change every 2 weeks. For the first 4 weeks of the study, participants will report via Interactive Voice Response (IVR) calls for 2 weeks and SMS text messages for 2 weeks. For the final two week period, research staff will help participants to set up the monitor to automatically send daily step counts to STEPS project staff. This can be done through a smartphone, tablet, or computer.
  Arms: STEPS Intervention Group

SUMMARY:
Wearable, commercially-available physical activity monitors are being increasingly incorporated into chronic pain self-management interventions as a tool to help patients set goals and to tailor intervention content based on patient progress. Yet older adults from resource-challenged communities may face significant barriers to using these monitors and reporting activity data. Our pilot study will focus on wearable monitor use among older adults in Detroit with chronic musculoskeletal pain, testing the feasibility and validity of various technology-based strategies for reporting daily step count data. The study will also assess whether six weeks of monitor use is associated with improvements in functioning, relative to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Ambulatory with or without assistive device
* Community living
* Have a SMS-capable cell phone
* Internet access (via smartphone, in-home or elsewhere);
* Self-reported chronic musculoskeletal pain (pain in muscles or joints for > 3 months)
* >4 (0-10 scale) average pain level over last week
* >1 day/previous 30 when pain made it difficult to do usual activities
* Ability to travel to study location in Detroit for a one-time session

Exclusion criteria:

* Serious acute illness or hospitalization in last month
* Planned surgery in next month
* Severe cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Janevic, Principal Investigator — University of Michigan School of Public Health
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant pre-assignment events.
Period: Overall Study
Arm/Group | STEPS Intervention Group | STEPS Control Group
Started | 33 | 24
Completed | 28 | 23
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not able to attend required orientation | 3 | 0

BASELINE CHARACTERISTICS:
Population: Note: This is the analytic sample (i.e., participants with baseline and 8-week follow-up data, representing 51 of 57 randomized.)
Groups:
- Total: Total of all reporting groups
Arm/Group | STEPS Intervention Group | STEPS Control Group | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (7.1) | 69.3 (6.4) | 70.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 21 | 48
  White | 0 | 0 | 0
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 23 | 51
Pain intensity in last week [Mean (Standard Deviation); unit: units on a scale] — Pain intensity rated on 1 to 10 scale, where 1=no pain and 10=worst imaginable pain).
  units on a scale | 5.1 (1.3) | 5.4 (2.2) | 5.2 (1.8)
PROMIS 4-item pain interference T-score [Mean (Standard Deviation); unit: units on a scale] — Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much). Converted to population-normed T-score (population mean of 50).
  units on a scale | 58.7 (6.1) | 57.0 (8.4) | 58.0 (7.2)
PROMIS 4-item physical function difficulty T-score [Mean (Standard Deviation); unit: units on a scale] — Items ask how much difficulty participant has in doing daily activities such as household chores, using stairs, and walking 15 minutes (1=without any difficulty to 5=unable to do). Converted to population-normed T-score (population mean of 50).
  units on a scale | 33.2 (4.3) | 31.9 (4.2) | 33.0 (5.2)
PROMIS 4-item social partcipation T-score [Mean (Standard Deviation); unit: units on a scale] — Items assess difficulty participating in family activities, leisure activities, and work 1=not at all to 5=very much). Converted to population-normed T-score (population mean of 50).
  units on a scale | 38.1 (7.3) | 37.0 (6.4) | 37.6 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Interference
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS-29) Pain Interference 4-item subscale, where a higher score indicates more pain interference. Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much). Raw scores are converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation). The possible range is 42 to 76, with a higher score representing worse outcome.
Time Frame: Baseline, eight weeks
Population: This is from the analytic sample that had both baseline and follow-up data on this measure. Change score is the follow-up minus baseline score, such that a greater, negative change value is a better outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEPS Intervention Group | STEPS Control Group
Number analyzed (Participants) | 28 | 23
score on a scale | -0.85 (6.2) | -0.21 (6.6)

2. Primary Outcome: Adherence to Step Count Reporting - SMS
Description: Proportion of days that step count was successfully provided/possible reporting days for SMS
Time Frame: Two weeks
Population: Intervention group participants with baseline and follow-up data. Excludes one case that did not have a texting plan on her phone. Result represents number of adherent person-days out of all possible person-days for SMS.
Measure: Count of Units; unit: person-days
Units Other Than Participants: person-days
Groups:
- STEPS Intervention Group: This analysis was only conducted on the Intervention group, who participated in 6 weeks of tracking and reporting step counts.
Arm/Group | STEPS Intervention Group
Number analyzed (Participants) | 27
Number analyzed (person-days) | 378
person-days | 299

3. Primary Outcome: Adherence to Step Count Reporting - IVR
Description: Proportion of days that step count was successfully provided/possible reporting days for IVR.
Time Frame: two weeks
Population: Intervention group participants with baseline and follow-up data. Excludes one case who did not receive IVR calls on schedule due to system error. Result represents number of adherent person-days out of all possible person-days for IVR.
Measure: Count of Units; unit: person-days
Units Other Than Participants: person-days
Arm/Group | STEPS Intervention Group
Number analyzed (Participants) | 27
Number analyzed (person-days) | 378
person-days | 257

4. Primary Outcome: Adherence to Step Count Reporting - Sync
Description: Proportion of days that step count was successfully provided/possible reporting days for syncing with app
Time Frame: two weeks
Population: Intervention group participants with baseline and follow-up data. Result represents number of adherent person-days out of all possible person-days for sync.
Measure: Count of Units; unit: person-days
Units Other Than Participants: person-days
Arm/Group | STEPS Intervention Group
Number analyzed (Participants) | 28
Number analyzed (person-days) | 392
person-days | 267

5. Secondary Outcome: Change in Physical Functioning
Description: The Physical Functioning 4-item subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Adult Profile. Items ask how much difficulty participant has in doing daily activities such as household chores, using stairs, and walking 15 minutes (1=without any difficulty to 5=unable to do); raw total scale scores range from 4 (high functioning) to 20 (low functioning). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 23 to 57, with a higher score representing worse outcome.
Time Frame: Baseline, eight weeks
Population: Participants who had data on both baseline and follow-up measure. Change score is the follow-up minus baseline score, such that a greater, negative change value is a better outcome.
Measure: Mean (Standard Deviation); unit: units on a scale (T-score)
Arm/Group | STEPS Intervention Group | STEPS Control Group
Number analyzed (Participants) | 28 | 23
units on a scale (T-score) | -1.4 (3.5) | -0.85 (3.7)

6. Secondary Outcome: Change in Social Participation
Description: Ability to Participate in Social Roles and Activities, a 4-item subscale from PROMIS-20 rating the amount of trouble (1=not at all to 5=very much) in participating in social roles such as family activities, leisure activities, and work. Raw total scale scores range from 4 (high functioning) to 20 (low functioning). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 29 to 64, with a higher score representing worse outcome.
Time Frame: Baseline, eight weeks
Population: Participants who had data on both baseline and follow-up measure. Change score is the follow-up minus baseline score, such that a greater, negative change value (or smaller positive value) is a better outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STEPS Intervention Group | STEPS Control Group
Number analyzed (Participants) | 28 | 23
units on a scale | 0.28 (7.8) | 0.83 (8.4)

7. Secondary Outcome: Validity of Manually-reported Step Count Data - SMS
Description: Correlation of manually-reported SMS data with automatically uploaded data - percentage of days that counts are within 50 steps of each other
Time Frame: Two weeks
Population: Result is number of person- days with valid data reported that were within 50 steps of sync value.
Measure: Count of Units; unit: person-days
Units Other Than Participants: person-days
Arm/Group | STEPS Intervention Group
Number analyzed (Participants) | 27
Number analyzed (person-days) | 256
person-days | 133

8. Secondary Outcome: Validity of Manually Reported Step Count Data - IVR
Description: as for outcome 7
Time Frame: Two weeks
Population: Result is number of person- days with valid data reported that were within 50 steps of sync value.
Measure: Count of Units; unit: person-days
Units Other Than Participants: person-days
Arm/Group | STEPS Intervention Group
Number analyzed (Participants) | 27
Number analyzed (person-days) | 215
person-days | 94

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | STEPS Intervention Group | STEPS Control Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STEPS Intervention Group (N=28) | STEPS Control Group (N=23)
hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant was hospitalized for pneumonia. Not related to research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03285958/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03285958/ICF_001.pdf